CLINICAL TRIAL: NCT06754111
Title: The Effect of Ideal Birth Environment on Birth Pain, Fear of Childbirth, Mode of Delivery and Duration of Delivery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Sema Göçmez, lecturer, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GO 2024/510
Record Dates: First submitted 2024-12-10; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Pregnant; Fear of Childbirth; Ideal Birth Environment
Keywords: labor pain; ideal birth environment; fear of childbirth
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): will receive standard care, no intervention will be performed
- ideal birth environment (Active Comparator): ideal birth room While designing a single room without unnecessary medical equipment, your own bed linen, bed linen, It will be a pillow case, a photo frame, he will be able to listen to the music he wants, he will be able to make a photo of his own choice.
  There will be a companion, a birthing ball and chair, and the room will allow freedom of movement.
  It will be designed to allow
  Interventions: Behavioral: ideal birth environment

INTERVENTIONS:
Behavioral: ideal birth environment — ideal birth room While designing a single room without unnecessary medical equipment, your own bed linen, bed linen, It will be a pillow case, a photo frame, he will be able to listen to the music he wants, he will be able to make a photo of his own choice.
  There will be a companion, a birthing ball and chair, and the room will allow freedom of movement.
  It will be designed to allow
  Arms: ideal birth environment

SUMMARY:
The aim of this study was to investigate whether the ideal birth environment is related to fear of childbirth, labor pain, duration of labor, and mode of delivery.

on the impact of the study. The main questions it aims to answer are Does the ideal birth environment reduce fear of childbirth? Does the ideal birth environment reduce labor pain? does the ideal birth environment affect the duration of labor? In order to evaluate the effect of the ideal birth environment on fear, pain and duration of labor, the researchers will compare the standard delivery room and women who will give birth in a room customized for women, where they have their own sheets, pillows, items that make them feel special, where medical devices are reduced, in a room where they have photos with their partner, in a room where they listen to the music they want, where they have freedom of movement. both in the experimental and control groups: In the last trimester, the Wijma birth experience A version will be applied and in the postpartum period, the Wijma B Birth experience scale will be applied again and the fear of childbirth will be evaluated. Pain in labor will also be assessed using VAS (Visceral Visual Analgesic Scale) during the latent and active phase of labor.

DETAILED DESCRIPTION:
The birth environment filled with medical instruments increases the level of anxiety and fear in the mother.

increase, disrupting the neurohormonal relationship that ensures the normal functioning of labor and an increase in the rate of cesarean section deliveries. Also women when she does not feel safe in her environment and her baby does not feel safe, the birth process is temporary. may slow down as a result release of adrenaline (epinephrine) and noradrenaline (norepinephrine) as a result of stress and anxiety increases, creating a "fight or flight" situation in the woman. Adrenaline and noradrenaline are the main

towards the end of labor to help the fetus to expel, while towards the end of labor should be at a low level at the beginning. The woman cannot fight stress in these cases, adrenaline and noradrenaline levels increase, while oxytocin levels decrease. This one from a physiological point of view, it can cause the progression of labor to stop, the duration prolonged labor and increased cesarean section rates. In a study conducted with pregnant rats, noise and movement in the birth environment restriction has been found to negatively affect hormones involved in labor

ELIGIBILITY:
Inclusion Criteria:

18-35 years old pregnant primiparous literate

Exclusion Criteria:

Medium and high-risk pregnant women (oligohydramnios, pre-eclampsia, heart disease, diabetes, placenta previa)

* Psychiatric illness such as anxiety and depression
* Communication barrier

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Wijma Birth Expectancy/Expectation Questionnaire (W-DEQ) A Version | 28-36 weeks of gestation
  Wijma Birth Expectancy/Expectation Scale A Version (W-DEQ A), W-DEQ consists of 33 items and is a six-point Likert-type scale.
  Item responses are numbered from 0 to 5, with 0 indicating "completely" and 5 indicating "not at all".
  is expressed. The minimum score is 0 and the maximum score is 165. The cut-off value is 85 points and a score of 85 and above is expressed as clinical fear.
  is also analyzed. The higher the total score of the scale, the higher the degree of fear experienced.
  is high.
  * W-DEQ score? 37 mild,
  * W-DEQ score = 38-65 moderate,
  * W-DEQ score = 66-84 in severe degree,
  * A W-DEQ score of ? 85 indicates a clinical degree of fear. Scale 2, Questions 3, 6, 7, 8, 11, 12, 15, 19, 20, 24, 25, 27 and 31 are negatively loaded and there is no agreement in the measurement.
  The alpha value of the scale is calculated by inverting the scale in the opposite direction. Cronbach's alpha value of the scale 0.89 (Korukcu et al., 2012) Wijma Birth Anticipation/Experience Sc
VASA Pain Assessment Scale | during the latent phase of labor when the cervical opening is 1-3 cm and during the active phase of labor when the cervical opening is 5-7 cm
  Quantitative pain rating scale (QPRS) is used to assess the severity of pain. is used. On a numerical rating scale, pain ranges from 0 (no pain) to 10 (unbearable pain) score (Price et al., 1983).
WIJMA BIRTH EXPECTANCY/EXPERIENCE SCALE B VERSION | up to the first 12 hours after birth
  he W-DEQ consists of 33 items and is a six-point Likert-type questionnaire. Item responses are numbered from 0 to 5, with 0 indicating "completely" and 5 indicating "not at all".
  is expressed. The minimum score is 0 and the maximum score is 165. The cut-off value is 85 points and a score of 85 and above is expressed as clinical fear.
  is also analyzed. The higher the total score of the scale, the higher the degree of fear experienced.
  is high.
  * W-DEQ score? 37 mild,
  * W-DEQ score = 38-65 moderate,
  * W-DEQ score = 66-84 in severe degree,
  * A W-DEQ score of ? 85 indicates a clinical degree of fear. Scale 2, Questions 3, 6, 7, 8, 11, 12, 15, 19, 20, 24, 25, 27 and 31 are negatively loaded and there is no agreement in the measurement.
  is calculated by inverting it in the opposite direction in order to provide
  Translated with www.DeepL.com/Translator (free version)

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Akif Ersoy Üniversitesi, Burdur, Bucak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No